CLINICAL TRIAL: NCT05068531
Title: A Prospective Observational Cohort Study for Early Detection of Treatment Failure in Metastatic Colorectal Cancer Patients Undergoing Systemic Chemotherapy and Liver Resection With Curative Intent
Brief Title: Early Detection of Treatment Failure in Metastatic Colorectal Cancer Patients
Acronym: eDetect-mCRC
Status: Recruiting | Type: Observational
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: 21.103
Record Dates: First submitted 2021-09-02; First posted 2021-10-06 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Real world data; Observational study; Circulating tumor DNA; Microbiome; Tumor immunology; Metastatic colorectal cancer; Liver metastasis; Biomarker
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Serial blood samples processed to obtain plasma for ctDNA and soluble factor research, buffy coat for genomic research, and mononuclear cells for live cells immune assays;
  * Tumor samples processed to allow genomic, proteomic and live cell research;
  * Adjacent non-tumoral tissue to allow genomic, proteomic and live cell research;
  * Stool samples at baseline and post neoadjuvant chemotherapy to allow metagenomics research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: We plan to recruit up to 100 mCRC patients with baseline resectable liver-restricted metastases (mCRC-LR) without evidence of extra-hepatic metastases, with primary tumor already or to be resected (metachronous or synchronous disease), planned to receive upfront FOLFOX-based preoperative neoadjuvant systemic chemotherapy, who achieved no-evidence of disease (NED) in the abdomen by standard imaging.

SUMMARY:
In North America, colorectal cancer patients with resectable liver-restricted metastases (mCRC-LR) are treated with approximately 6 months of preoperative systemic multi-agent chemotherapy. Actuarial data however supports that approximately 20% of mCRC-LR patients can be cured without as much systemic chemotherapy. Prospective phase II-III trials also support that awaiting recurrence to initiate further metastases-targeted or systemic treatment may provide patients with longer overall survival while avoiding toxicities in those without recurrence.

DETAILED DESCRIPTION:
The general objective of this single-centre, prospective observational cohort study in 100 mCRC-LR patients treated with curative intent along standard of care (SOC), is to obtain real-world data on administered therapies, selected complications, and oncological outcomes, while longitudinally collecting biospecimens to enable correlative research investigating early biological markers of treatment resistance and recurrence.

Cryopreservation of sequential blood derivatives, tumor tissue, and stool samples will allow investigation of circulating tumor DNA (ctDNA), T-cell receptor repertoire, somatic cancer mutations, immune and other gene expression, gut microbiome, and soluble factors.

The first biological marker that will be investigated in correlative research will be longitudinal measurements of ctDNA targeting 30 oncogenes, 23 axons, and 146 hotspots (Follow It assay, Canexia Health). Additional biological markers will be defined in subsequent amendments to this protocol.

The results are expected to provide important insights for the design of future trials investigating ways to personalize therapy, such as to: a) avoid the unnecessary use of neoadjuvant or adjuvant systemic chemotherapy, b) avoid morbid hepatectomies in patients unlikely to benefit, c) test novel preoperative therapies in patients more likely to benefit, and d) modulate the intensity of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients (≥18 years of age at the time of consent);
2. Stage IV colon or rectal adenocarcinoma with liver-restricted metastasis(es) for whom partial hepatectomy with curative intent is planned;
3. Instead of, or in addition to, partial hepatectomy, liver metastases may be ablated by needle radio frequency or microwave; in case of a solitary liver metastasis, three core-needle biopsies are provided for research at time of the procedure and prior to tissue destruction;
4. Patients may undergo planned two-stage partial hepatectomies;
5. Patients may have at baseline lung micro nodules or intra-abdominal enlarged nodes or nodules of unknown nature, not considered as extra-hepatic metastases in the opinion of the investigator;
6. Patients who are scheduled to receive FOLFOX-based pre-hepatectomy may receive any additional combined agents, such as and not limited to Irinotecan, anti-EGFR, and anti-VEGF drugs;
7. Patients are willing and able to provide serial blood samples, tumor and adjacent tissues, and stool samples for research;
8. The timing and specific treatments of the primary colon or rectal tumor is per SOC, at the discretion of the treating physician, including the use of pre-operative radiotherapy for rectal cancer;
9. Patients may receive post-operative adjuvant chemotherapy per SOC, at the discretion of the treating physician;
10. Patients must consent to the Exactis Personalized my Treatment registry.

Exclusion Criteria:

1. Pregnant or breastfeeding patients,
2. Hereditary colorectal cancer (e.g., familial colonic polyposis or Lynch syndrome), and
3. Presence of concurrent other cancer(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 100 mCRC patients with baseline resectable liver-restricted metastases (mCRC-LR) without evidence of extra-hepatic metastases, with primary tumor already or to be resected (metachronous or synchronous disease), planned to receive upfront FOLFOX-based preoperative neoadjuvant systemic chemotherapy, who achieved no-evidence of disease (NED) in the abdomen by standard imaging.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Radiological response to pre-operative chemotherapy as assessed by RECIST v1.1 | Approximately three months
Biochemical response to pre-operative chemotherapy as assessed by plasmatic CEA measurement, change from baseline after 4 cycles of chemotherapy | Approximately three months
Pathological response to pre-operative chemotherapy as assessed by Ryan and Rubbia Brandt Tumor Regression Grade (TRG) scores on resected tumors | Approximately three months
Tumor response to pre-operative chemotherapy as assessed by change in circulating tumor DNA level, change from baseline | Approximately three months
  Follow It assay, Canexia Health
Histopathologic growth pattern as assessed by percent replacement, desmoplastic, and pushing features measured at the interface of liver metastasis and non tumoral liver | Three to four months
Post-operative minimal residual disease as assessed by circulating tumor DNA detection after tumor resection with curative intent | Approximately 1 months after resection with curative intent
  Follow It assay, Canexia Health
Time to radiological recurrence after tumor resection with curative intent | Up to three years after tumor resection with curative intent
Time to biochemical recurrence as assessed by plasmatic CEA measurement, level above the upper limit occurring after tumor resection with curative intent | Up to three years after tumor resection with curative intent
Time to tumor recurrence as assessed by detection or change in level of circulating tumor DNA after tumor resection with curative intent | Up to three years after tumor resection with curative intent
  Follow It assay, Canexia Health

SECONDARY OUTCOMES:
Incidence and grade of FOLFOX-induced neuropathy, as assessed by Sensory Subscale of the NCI CTCAE scale, version 3 | Two to three months pre-operatively and during post-operative adjuvant chemotherapy
Incidence of allergic reaction to oxaliplatin diagnosed by treating physicians and requiring desensitization or change in chemotherapy regimen | Two to three months pre-operatively and during post-operative adjuvant chemotherapy
Incidence of hospitalization for febrile neutropenia diagnosed by treating physicians | Two to three months pre-operatively and during post-operative adjuvant chemotherapy
Ninety-day post-surgical complications, defined by Clavien Dindo grading system | 90 days after tumor resection
Disease-specific survival after complete tumor resection | Up to three years after tumor resection with curative intent

CONTACTS AND LOCATIONS:
Overall Officials: Simon Turcotte, MD, MSc, Principal Investigator — CHUM
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided